CLINICAL TRIAL: NCT06606561
Title: A Phase I/II Randomized, Double Blinded, Placebo Controlled Trial to Evaluate the Safety and Potential Efficacy of NANOVAE Injected Intra-Articular in Patients Suffering With Knee Osteoarthritis
Brief Title: NANOVAE to Treat Knee Osteoarthritis (KOA)
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nova Vita Laboratory (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NVL-2024-257
Record Dates: First submitted 2024-09-17; First posted 2024-09-23 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A total of 24 subjects meeting all inclusion/exclusion criteria will be divided into two groups. Group 1 will be an open-label lead-in phase. Group 2 will be a randomized, double-blinded, placebo-controlled cohort. Group 1 will receive one dose of 2ml of NANOVAE, and Group 2, in a randomized and double-blinded fashion, will receive two doses of 2ml NANOVAE. Neither the patients nor the researchers will know who is getting the placebo and who is getting the NANOVAE; only the product manufacturing staff will be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Open Label) (Experimental): A total of eight subjects will be treated to assess safety prior to enrolling Group 2. We propose to assess the safety of 8 subjects in Group 1 at seven-day intervals. Each subject in Group 1 will be staggered by 5 days after receiving the dose of NANOVAE.
  Dose - 2 mL of NANOVAE on day 0 containing 1.0 x 1011 to 9.0 x 1011 particles/ml. Product will be administered directly without any dilution.
  Interventions: Drug: NANOVAE - Acellular Allogenic Human Amniotic Fluid (hAF)
- Group 2 (Randomized, double blinded placebo control) (Experimental): Total of sixteen subjects will be randomized to either receive two doses of NANOVAE via intraarticular injections or receive two doses of a placebo.
  Dose - 2 mL of NANOVAE or placebo on day 0 and day 15, containing 1 x 1011 particles/ml. The ratio is 1:1 for a total of 16 subjects in the Group 2. Product will be administered directly without any dilution.
  Interventions: Drug: NANOVAE - Acellular Allogenic Human Amniotic Fluid (hAF); Drug: 0.9% Sodium Chloride Injection, USP

INTERVENTIONS:
Drug: NANOVAE - Acellular Allogenic Human Amniotic Fluid (hAF) — A total of 24 subjects meeting all inclusion/exclusion criteria will be divided into two groups. Group 1 will be an open-label lead-in phase. Group 2 will be a randomized, double-blinded, placebo-controlled cohort. Group 1 will receive one dose of 2ml of NANOVAE, and Group 2, in a randomized and double-blinded fashion, will receive two doses of 2ml NANOVAE. Neither the patients nor the researchers will know who is getting the placebo and who is getting the NANOVAE; only the product manufacturing staff will be unblinded. The ratio of placebo to NANOVAE is 1:1 for a total of 16 subjects in Group 2. Only the knee with the more severe symptoms of OA will be treated. The allogenic-HAF
Drug: 0.9% Sodium Chloride Injection, USP — In lieu of AF, the saline for injection will be used as a placebo. Vials acquired from the manufacturer is pipetted into glass vials, stoppered, capped, placed in labeled header foil pouches, and sealed. These are transferred to a quarantine freezer to await post-production testing.
  Other Names: Placebo
  Arms: Group 2 (Randomized, double blinded placebo control)

SUMMARY:
The below summarizes relevant information for investigator(s) to consider the use of Allogenic Human Amniotic Fluid product in a clinical protocol detailing study design and conduct for a phase I/II randomized, double-blinded, placebo-controlled clinical trial to evaluate the safety and potential efficacy of NANOVAE injected intra-articularly in patients suffering from knee osteoarthritis. The IB will be reviewed annually and amended when further information becomes available.

Osteoarthritis (OA) is a degenerative disease of the joints that affects millions of people worldwide, yet its exact causes are not fully understood. Middle-aged to elderly individuals are often the most impacted by OA, which primarily affects the knee, hip, spine, and joints in the fingers. Among these, knee osteoarthritis (KOA) is the most common form, causing pain, stiffness, and reduced functionality, and it is a major contributor to chronic bone and muscle pain. It is also a leading cause of disability in adults who are not living in institutions. Treatment for KOA is challenging due to its resistance to medications, procedures, and surgeries. The primary objective is to alleviate pain and enhance overall function. However, since there is currently no cure for OA, the need for an effective therapy remains urgent. Healthcare professionals often encounter patients whose pain may result from an inflammatory response triggered by injury or disease. Research suggests that regenerative medicine, utilizing techniques like stem cells, platelet-rich plasma (PRP), amniotic fluid, and cytokine modulation, holds promise for treating KOA.

OA is associated with an increase in pro-inflammatory substances such as interleukin (IL)-1, IL-6, tumor necrosis factor-alpha (TNF-α), matrix metalloproteinases (MMPs), nitric oxide (NO), reactive oxygen species (ROS), and cytokine-inducible cyclooxygenase-2 (COX-2). These inflammatory agents affect various cell types within the affected joints, including chondrocytes, osteoblasts, osteoclasts, synoviocytes, and macrophages. Some miRNAs, which are downregulated in OA, have been identified as protective factors. For example, miR-130 helps regulate TNF-α levels, while miR-149 controls several inflammatory cytokines such as IL-1, IL-6, and TNF-α. The breakdown of the cartilage matrix is a key characteristic of OA. MMP-13, a member of the MMP family, plays a significant role in degrading the collagen network during OA development. Several miRNAs, including miR-27b, miR-27a, miR-148a, miR-320, miR-127-5p, and miR-411, are downregulated in OA and target the mRNA of this proteinase. It is important to note that a single miRNA can regulate multiple target genes associated with OA progression. For instance, miR-105 and miR-148, both downregulated in OA, target genes such as Runx2, ADAMTS4, ADAMTS5, ADAMTS7, ADAMTS12, MMP-13, and COL10, implying their potential protective roles.

Several studies have shown a link between certain miRNAs, aging, and the progression of OA. For example, miR-320c is downregulated in aging OA samples and regulates ADAMTS5, suggesting that this miRNA may serve as a protective factor by enhancing chondrogenesis.

DETAILED DESCRIPTION:
The investigational product being assessed in this trial is called NANOVAE, which is a biologic derived from human amniotic fluid (HAF) that is allogenic and acellular. HAF contains a wide range of growth factors, cytokines, chemokines, and extracellular vesicles/nanoparticles obtained from perinatal tissue. These components contribute to the regenerative potential of HAF and make it a promising option for regenerative medicine applications, particularly in knee osteoarthritis (KOA). Studies have demonstrated that the extracellular vesicles found in HAF, including exosomes, have the ability to promote chondrogenesis and reduce inflammation, which are crucial processes in reversing the progression of KOA. Additionally, these vesicles have shown to stimulate cartilage regeneration, addressing the impaired cartilage repair typically observed in OA. Therefore, the administration of HAF-derived products has the potential to slow down the degenerative process and promote cartilage repair in patients with KOA. The growth factors and cytokines present in HAF may also help alleviate the inflammatory response observed in the knee joint, a characteristic feature of KOA. These anti-inflammatory properties, combined with the regenerative capabilities of the extracellular vesicles, make HAF an appealing candidate for the treatment of KOA.

Numerous clinical studies registered under ClinicalTrials.gov have provided evidence of the safety and effectiveness of HAF products in joint therapies. The use of HAF for treating OA holds immense potential due to its array of growth factors, anti-inflammatory mediators, and medicinal signaling cells, which continue to undergo rapid advancements. In a non-FDA review study, a double-blinded controlled trial was conducted comparing the treatment of OA with freshly collected amniotic fluid and steroids. The results revealed a significant improvement in the Visual Analog Scale (VAS) after three months of treatment, with continuous improvement in VAS after six months in both groups. However, the group receiving freshly collected amniotic fluid exhibited greater improvement. These findings strongly support the potential of this novel HAF therapy for advanced OA, as it proved to be superior and longer lasting compared to conventional therapies commonly practiced. Further research, both in terms of basic science and clinical investigations, is warranted to gain a better understanding of the anti-inflammatory properties of amniotic fluid and determine the most efficacious amniotic fluid product for symptomatic OA.

NANOVAE is a filtered form of HAF (human amniotic fluid) that utilizes the wide range of nanoparticles, cytokines, and growth factors present in the fluid, which play vital roles in fetal development and maturation. HAF is a rich source of collagen substrates, growth factors, amino acids, polyamines, lipids, carbohydrates, cytokines, and extracellular matrix molecules like hyaluronic acid and fibronectin, as well as cells. These components greatly contribute to tissue protection and repair. Extensive research has demonstrated the antimicrobial, immunomodulatory, and growth-promoting properties of HAF. The antimicrobial, antiviral, and antifungal effects of HAF have been established through the identification of various components such as lysozyme, peroxidase, transferrin, β-lysin, immunoglobulins, and zinc-peptide complexes within the fluid. The immunomodulatory functions of HAF have been observed in its ability to suppress alloreactive responses and downregulate Th1 and Th2 cytokines.

NANOVAE's extracellular vesicle (EV) fraction consists of several cytokines, chemokines, and growth factors that are associated with functions such as host defense, anti-inflammatory response, angiogenesis, and cartilage repair. The concentration of nanoparticles in the final product has been consistently demonstrated through nanoparticle analysis using the ZetaView Quatt nanoparticle analyzer. This analysis reveals a range of particles, with an average mode particle size of 96.4 nM, which aligns with the expected size of exosomes ranging between 50-200 nm in diameter.

Objectives:

Primary Objective: To demonstrate the safety of NANOVAE administered intraarticular in subjects with KOA by measuring the incidence of any of the following treatment-emergent adverse events (TE-AEs) and treatment-emergent serious adverse events (TE-SAEs) within the first 30 days of injection:

Occurrence of adverse events related to the therapy within 30 days of NANOVAE treatment.

Life-threatening event (e.g., stroke or non-fatal pulmonary embolism). Event resulting in persistent or significant disability/incapacity. Event resulting in death.

Secondary Objective: To demonstrate the potential efficacy of NANOVAE by measuring the following clinical response changes from baseline to 12 months after injection. Time Frame: Month 1, 3, 6, and 12 after infusions:

Change in single leg stance test. Change in "Timed Up and Go" test to assess fall risk. Change in Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index (five items for pain, two for stiffness, and seventeen for function).

Change in range of motion, assessed by goniometer measurements. Change in serum and/or synovial biomarkers between the timepoints of Day 0 and the 3-month visit.

Design and Investigational Plan: A total of 24 subjects meeting all inclusion/exclusion criteria will be divided into two groups. Group 1 will be an open-label lead-in phase. Group 2 will be a randomized, double-blinded, placebo-controlled cohort. Group 1 will receive one dose of 2ml of NANOVAE, and Group 2, in a randomized and double-blinded fashion, will receive two doses of 2ml NANOVAE. Neither the patients nor the researchers will know who is getting the placebo and who is getting the NANOVAE; only the product manufacturing staff will be unblinded. The ratio of placebo to NANOVAE is 1:1 for a total of 16 subjects in Group 2. Only the knee with the more severe symptoms of OA will be treated. The allogenic-HAF will be obtained from healthy donors and manufactured by the Nova Vita Laboratories processing lab.

Group 1 (Open Label): A total of eight subjects will be treated to assess safety prior to enrolling Group 2. Safety will be assessed at seven-day intervals for the 8 subjects in Group 1, staggered by 5 days after receiving the dose of NANOVAE.

Dose: 2 mL of NANOVAE on Day 0 containing 1.0 x 10¹¹ to 9.0 x 10¹¹ particles/ml. Product will be administered directly without any dilution.

After these 8 subjects complete the 5-day safety assessment, the safety report will be presented to the DSMB with representative data to determine the safety status of receiving one dose of NANOVAE. Once the treatment of Group 1 has been determined to be safe, the enrollment of Group 2 will begin.

Group 2 (Randomized, double-blinded placebo control): A total of sixteen subjects will be randomized to either receive two doses of NANOVAE via intraarticular injections or receive two doses of a placebo.

Dose: 2 mL of NANOVAE or placebo on Day 0 and Day 15, containing 1 x 10¹¹ particles/ml. The ratio is 1:1 for a total of 16 subjects in Group 2. Product will be administered directly without any dilution.

Sample Size & Study Population: A total of 24 adult patients will be chosen from the population of adults between the ages of 21 to 75 diagnosed with KOA who meet inclusion criteria.

Route of Administration: Intra-articular Injections.

Study Duration and Study Follow-Up: 12 months total duration:

Day 0 and 15 - Intraarticular Injection and observational follow-up. Days 1 and 7 (after dose of NANOVAE or placebo) - Observational follow-up via phone call, telehealth, or in-person visit.

Months 1, 3, 6, and 12 - Observational follow-up visits per protocol design.

ELIGIBILITY:
Inclusion Criteria:

1. Age eligible for study: 21 to 75 years
2. Gender eligible for study: All
3. Study subjects must be willing to give written informed consent to participate in the study and sign the Health Insurance Portability and Accountability Act (HIPAA) authorization before any study procedures are performed.
4. Subjects have a diagnosis of OA in at least one knee defined as Grade II or III on Kellgren-Lawrence (K-L) grading scale which is confirmed by posterior-anterior, weight-bearing, fixed flexion radiography with 10o caudal beam angulation.
5. Subjects with VAS pain score ≥40 mm on screening day will be included.
6. Subjects had one or more of the following SOC treatments within the previous 12 months will be included:

   1. weight loss
   2. physical therapy
   3. anti-inflammatory medications - oral, injections and topical
7. Body mass index (BMI) < 45kg/m2
8. Subjects must be available for all specified assessments at the study site through the completion of the study.
9. For Women of Child-Bearing Potential (WOCBP) only, willingness to use FDA-recommended birth control until 6 months post treatment. The FDA-approved and cleared methods for birth control are listed below:

   1. Permanent Sterilization
   2. Long-Acting Reversible Contraceptives (LARC)
   3. Contraceptive Injection
   4. Short-Acting Hormonal Methods
   5. Barrier Methods
   6. Emergency Contraception https://www.fda.gov/consumers/free-publications-women/birth-control
10. Any male subject must agree to use contraceptives and not donate sperm during the study.
11. Patient may be eligible for treatment of both knees if criteria is met for both

Exclusion Criteria:

1. Subjects have evidence of significant and unstable cardiac dysfunction, e.g. acute myocardial infarction and hypertension with uncontrolled blood pressure over 140/90 will be excluded.
2. Subjects at screening with white blood cell count < 4 x 109 cells/L, hematocrit <30%, and platelets <150 x 109 /L will be excluded.
3. Subjects with poorly controlled diabetes (hemoglobin A1C > 7.5 or fasting blood glucose of >200) in last 6 months will be excluded.
4. Individuals on dialysis or uncontrolled renal disease will be excluded.
5. Subjects with abnormal hematology, serum chemistry, or urinalysis screening laboratory results will be excluded.
6. Subjects with history of, or ongoing, autoimmune disorder that requires treatment with an immunosuppressive medication will be excluded.
7. Subjects had knee surgery on the targeted knee within 12 months prior to screening and /or planned knee surgery during the study will be excluded.
8. Subjects have a body mass index greater than 45 kg/m2 will be excluded.
9. Subjects whose knee pain is caused by, (i) diffuse edema, extra articular causation (ii) displaced meniscus tear, (iii) full thickness articular cartilage lesion greater than 1 cm in any direction, or (iv) osteochondritis dissecans will be excluded.
10. Subjects have rheumatoid arthritis, psoriatic arthritis, or have been diagnosed with any other auto-immune disorders that could be the cause of their knee pain will be excluded.
11. Subjects which have evidence or history of malignancy except those who are successfully treated in situ or basal cell skin cancers will not be excluded.
12. Subjects with a history of clotting disorder, anticoagulation therapy that cannot be stopped as prior to infusion will be excluded.
13. Subjects have evidence of liver dysfunction manifested as alkaline phosphatase greater than 345 u/L, total bilirubin greater than 1.65 mg/dL, ALT greater than 275 units/L and/or AST great than 240 units/L will be excluded.
14. Subjects have or had an active infection requiring systemic antibiotics within 2 weeks on enrollment in the study will be excluded.
15. Subjects currently taking anticoagulant therapy (excluding Plavix or Aspirin) will be excluded.
16. Subjects have received an intra-articular hyaluronic acid (HA) or platelet rich plasma (PRP) for the treatment of OA of the target knee within 12 weeks prior to screening will be excluded.
17. Subjects have used an investigational drug or had surgical intervention within 12 weeks of the study enrollment will be excluded.
18. Subjects that are unwilling to stop taking prescription or over the counter pain medication for Osteoarthritis for 7 days prior to any visit will be excluded. Subjects will be permitted to take medications for non-osteoarthritis condition (excluding the one's listed under "Concomitant Medication").
19. Subjects needing or at high risk of requiring systemic steroids during the course of study will be excluded except systemic use of corticosteroid administration for COVID-19 or flare up of non-arthritic condition.

    Complete information of dose and timeframe of the medication use will be documented in case report forms (CRF).
20. Be a female who is pregnant, nursing, or of childbearing potential while not practicing effective contraceptive methods.
21. Subjects who are unable to complete all the testing required for the study will be excluded.
22. Subjects on active listing (or expected future listing) for transplant of any organ will be excluded.
23. Be a solid organ transplant recipient. This does not include prior cell-based therapy (>12 months prior to enrollment), bone, skin, ligament, tendon or corneal grafting. Have a history of organ or cell transplant rejection.
24. Subjects with history of drug abuse (illegal "street" drugs except marijuana (If it is legal use in states where patient resides), or prescription medications not being used appropriately for a pre-existing medical condition or alcohol abuse (≥ 5 drinks/day for ˃ 3 months).
25. Subjects with untreated HIV infection will be excluded. However, patients can be enrolled if have been treated for HIV and the test negative for HIV viral load but still test positive for antibodies.
26. Subjects with neural or vascular claudication or neurologic disorder including, but not limited to epilepsy, Parkinson's disease, dementia, cerebrovascular disease, tumor of the nervous system, and amyotrophic lateral sclerosis will be excluded.
27. Subjects cannot have had a hyaluronic acid injection within 6 months prior to NANOVAE injection
28. Subjects cannot have had a cortisone injection within 3 months prior to NANOVAE Injection

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of NANOVAE administered intraarticular in subjects | 30 Days
  To demonstrate the safety of NANOVAE administered intraarticular in subjects with KOA by measuring incidence of any of the following treatment-emergent adverse events (TE-AEs) and treatment-emergent serious adverse events (TE-SAEs) within the first 30 days of injection:
  * Occurrence of adverse events related to the therapy within 30 days of NANOVAE treatment.
  * Life-threatening event (e.g., stroke or non-fatal pulmonary embolism).
  * Event resulting in persistent or significant disability/incapacity.
  * Event resulting in death.

SECONDARY OUTCOMES:
Change in Single Leg Stance Test | Baseline, Month 1, 3, 6, and 12 after infusions
  The Single Leg Stance Test will measure the ability of participants to balance on one leg for a specified duration. The test will be performed with eyes open and closed, and the time participants can maintain balance on a single leg without support will be recorded in seconds. The minimum value is 0 seconds, indicating inability to balance, and there is no fixed maximum value. Higher values indicate a better outcome (i.e., improved balance).
Change in "Timed Up and Go" Test | Baseline, Month 1, 3, 6, and 12 after infusions
  The Timed Up and Go (TUG) Test will assess participants' mobility and fall risk by measuring the time (in seconds) taken to stand up from a seated position, walk a short distance (approximately 3 meters), turn around, walk back to the chair, and sit down. The test will be timed using a stopwatch. The minimum time is 0 seconds, and no fixed maximum time is specified. Lower values indicate a better outcome (i.e., faster and safer mobility).
Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Baseline, Month 1, 3, 6, and 12 after infusions
  The WOMAC Index will be used to assess the participants' pain, stiffness, and physical function. It includes 5 items for pain, 2 for stiffness, and 17 for function, each rated on a scale of 0 to 4 (0 = none, 4 = extreme). The minimum total score is 0, and the maximum total score is 96. Higher scores indicate a worse outcome, meaning increased pain, stiffness, and dysfunction.
Change in Serum and/or Synovial Biomarkers | Baseline, Month 1, 3, 6, and 12 after infusions
  This outcome will track changes in serum and/or synovial fluid biomarkers relevant to inflammation and cartilage degradation. Biomarkers such as interleukin-1 (IL-1), tumor necrosis factor-alpha (TNF-α), and matrix metalloproteinases (MMPs) will be measured at baseline and at the 3-month visit. The results will be reported as concentrations (e.g., pg/mL or ng/mL), with lower levels of inflammatory biomarkers indicating a better outcome.
Change in Range of Motion (ROM) | Baseline, Month 1, 3, 6, and 12 after infusions
  Range of Motion will be measured using a goniometer to assess the degree of flexibility and movement in the knee joint. The test will measure both flexion and extension angles in degrees. The minimum ROM is 0 degrees (indicating no movement), and the maximum depends on the individual's ability. Higher values indicate a better outcome (i.e., increased mobility).

CONTACTS AND LOCATIONS:
Locations (1):
- Bluetail Medical Group, Chesterfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kohn MD, Sassoon AA, Fernando ND. Classifications in Brief: Kellgren-Lawrence Classification of Osteoarthritis. Clin Orthop Relat Res. 2016 Aug;474(8):1886-93. doi: 10.1007/s11999-016-4732-4. Epub 2016 Feb 12. No abstract available. PMID 26872913